CLINICAL TRIAL: NCT05695807
Title: Efficacy of Carboxy Therapy Versus Fractional Laser CO2 Versus Platelet Rich Plasma in Atrophic Scars, a Comparative Study.
Brief Title: Carboxytherapy in the Treatment of Atrophic Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Carboxytherapy atrophic scar
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Atrophic Scar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carboxytherapy (Experimental): Device
  Interventions: Device: Carboxytherapy
- Fractional CO2 laser (Active Comparator): Device
  Interventions: Device: Carboxytherapy
- Platelet rich plasma (Active Comparator): platelet rich plasma
  Interventions: Device: Carboxytherapy

INTERVENTIONS:
Device: Carboxytherapy — Device generating CO2 gas

SUMMARY:
To evaluate the efficacy of CO2 versus fractional CO2 laser versus platelet rich plasma in treatment of atrophic scars using clinical assessment and ultrasonography

ELIGIBILITY:
Inclusion Criteria:

* traumatic and surgical scar

Exclusion Criteria:

* active infections

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Modified Vancouver score | 12 weeks